CLINICAL TRIAL: NCT04145817
Title: Clinical Application of the European Horizon 2020 Research Project "BRIDGES" - Study of the Psychological Impact of Breast Cancer Risk Communication in Cancer Genetics Based on the Personalized Estimation of the BOADICEA V5/PLUS Model
Brief Title: Breast Cancer Risk After Diagnostic Gene Sequencing
Acronym: BRIDGEScohort2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IC 2018-08
Record Dates: First submitted 2019-07-18; First posted 2019-10-31 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Genetic Predisposition to Disease
Keywords: Related women to index case; Risk estimation; Breast cancer; Ovarian cancer
MeSH Terms: conditions — Genetic Predisposition to Disease; Breast Neoplasms; Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Women referred to genetic counselling in the participating Cancer Genetic Clinics will be included according to the selection criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- genetic counselling (Experimental): Genetic counselling (PRS for risk estimation) and questionnaires in the participating Cancer Genetic Clinics for healthy woman relative of a person first tested in the family (index case) who received a positive genetic test result or a negative non-informative test result
  Interventions: Genetic: BRIDGES gene panel testing; Genetic: Breast cancer risk polygenic risk score (PRS); Behavioral: Questionnaires

INTERVENTIONS:
Genetic: BRIDGES gene panel testing — The "Breast and Ovarian Analysis of Disease Incidence and Carrier Estimation Algorithm-BOADICEAV5/PLUS" predicts lifetime and age-specific breast cancer (BC) risks on the basis of family history, all known BC genes test-results, common single nucleotide polymorphisms (SNPs) combined in a PRS, and other non-genetic risk factors. This model is developed within the BRIDGES consortium.
Genetic: Breast cancer risk polygenic risk score (PRS) — The "Breast and Ovarian Analysis of Disease Incidence and Carrier Estimation Algorithm-BOADICEAV5/PLUS" predicts lifetime and age-specific breast cancer (BC) risks on the basis of family history, all known BC genes test-results, common single nucleotide polymorphisms (SNPs) combined in a PRS, and other non-genetic risk factors. This model is developed within the BRIDGES consortium.
Behavioral: Questionnaires — Self-administered questionnaires for counselees to evaluate Psychosocial Aspects of Hereditary Cancer (PAHC), Breast Cancer risk perception adequacy, risk communication within the family and cancer risk management choice,

SUMMARY:
Study of the psychological impact of breast cancer risk communication in Cancer Genetics based on the personalized estimation of the BOADICEA V5/PLUS model ("Breast and Ovarian Analysis of Disease Incidence and Carrier Estimation Algorithm-version 5 or PLUS").

DETAILED DESCRIPTION:
The new BC gene testing and risk estimation using BOADICEA V5/PLUS model imply an increased complexity of communication during the cancer genetic consultation. It will be proposed to women referred to genetic counselling in the participating Cancer Genetic Clinics .

New qualitative (moderate risks, secondary results) and quantitative results (variation in the degree of cancer risk identified for the counselee and family members) and thus a personalized breast cancer risk may be obtained. How this complexity affects counselees' psychological reactions is not known.

It is primarily aimed at comparing psychosocial needs and distress in healthy women (unaffected with BC) at high risk of breast or ovarian cancer undergoing genetic testing based on an enriched gene panel (index case gene panel plus PRS) at Curie Institute in France and at the University Hospital in Cologne, Germany.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy woman, relative of a family member first tested (index case) who received a positive genetic test result (presence of a BRCA1 or BRCA2 deleterious variant or a moderate-penetrance BC gene deleterious variant) ;

   a. at Cologne University Hospital (Germany), these healthy women may also be relatives of women (index case) who received a negative non-informative test result;
2. Who accept BRIDGES gene panel testing and the breast cancer risk PRS;
3. Aged 18 years or over with no upper limit;
4. Able to give informed written consent in accordance with national/local regulations and procedures;
5. Able to understand the questionnaire language of the participating genetic clinic.

Exclusion Criteria:

1. Woman affected with BC, with recurrent BC, with metastatic BC, with an ovarian cancer (OC) or cancer of any other site;
2. Aged under 18 years old;
3. Unable to give informed written consent;
4. Unable to understand the questionnaire language of the participating clinic;
5. Unable to answer the questionnaire due to physical or cognitive disturbance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 405 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Psychosocial Assessment in Hereditary Cancer questionnaire (PAHC). | Up to 6 months
  Breast or ovarian cancer risk perception (the impact of communicating a personalized breast cancer risk using the BOADICEAV5/PLUS model) using a PAHC questionnaire. Questionnaire items are responded on a 4-level scale from 1 (Not at all) to 4 (Very much). Item response scores are averaged and standardized on a 0 to 100 scale, with an increased value indication more severe difficulties.

SECONDARY OUTCOMES:
Difference on the PAHC score between counselees who receive a pathogenic variant indicating breast cancer versus (VS) who did not receive such result | Up to 6 months
  Counselee's perceived lifetime risks of developing (a first or second) BC will be measured at T2 in words (Not concerned, Don't know, Low risk, Low to moderate risk, Moderate risk, High risk, Very high risk, Major Risk) and in figures (Not concerned, Don't know, 0-10%; between 11-20%, 21-40%, 41-60%, 61-80% and over 80%).
Percentage of counselees intending to undertake risk reducing mastectomy (the one who received a pathogenic variant VS who did not receive such result) | Up to 6 months
  Counselees' choice of cancer risk management will be assessed using a study-specific self-administered questionnaire based on the literature [Julian-Reynier, 2010] asking about women's intention or choice to undergo regular mammography, regular breast ultrasound, MRI or preventive mastectomy on a 6-option response scale (Yes, certainly; Yes, probably; I don't know; No, probably not; No, certainly not; Not concerned).
Percentage of counselees who communicate their result to their sister(s) (the one who received a pathogenic variant VS who did not receive such result) | Up to 6 months
  It will be assessed using a study-specific self-administered questionnaire based on the literature [de Geus, 2015] asking about women's whether they informed about genetic testing among her husband/partner, children, mother, father, sister(s), brother(s), friend(s) or other family member(s) using a 4, 5 or 5-option response scale depending on the person (Yes, I informed him/her/them; No, but I plan to do it; No (no partner); No; Yes all of them; Yes, some of them; No (children too young); No (no children/brother/sister); No (mother/father deceased).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FUMOLEAU, MD, Study Chair — Institut Curie
Locations (2):
- Institut Curie, Paris, France
- University Hospital of Cologne, Cologne, Germany

REFERENCES:
- [Result] Bredart A, De Pauw A, Tuchler A, Lakeman IMM, Anota A, Rhiem K, Schmutzler R, van Asperen CJ, Devilee P, Stoppa-Lyonnet D, Kop JL, Dolbeault S. Genetic clinicians' confidence in BOADICEA comprehensive breast cancer risk estimates and counselees' psychosocial outcomes: A prospective study. Clin Genet. 2022 Jul;102(1):30-39. doi: 10.1111/cge.14147. Epub 2022 May 16. PMID 35508697
- [Result] Bredart A, Kop JL, Tuchler A, De Pauw A, Cano A, Dick J, Rhiem K, Devilee P, Schmutzler R, Stoppa-Lyonnet D, Dolbeault S. Assessment of psychosocial difficulties by genetic clinicians and distress in women at high risk of breast cancer: a prospective study. Eur J Hum Genet. 2022 Sep;30(9):1067-1075. doi: 10.1038/s41431-022-01096-9. Epub 2022 Apr 11. PMID 35399119
- [Result] Bredart A, De Pauw A, Anota A, Tuchler A, Dick J, Muller A, Kop JL, Rhiem K, Schmutzler R, Devilee P, Stoppa-Lyonnet D, Dolbeault S. Information needs on breast cancer genetic and non-genetic risk factors in relatives of women with a BRCA1/2 or PALB2 pathogenic variant. Breast. 2021 Dec;60:38-44. doi: 10.1016/j.breast.2021.08.011. Epub 2021 Aug 23. PMID 34455229